CLINICAL TRIAL: NCT00494013
Title: Treat-to-Target Comparison of Two Basal Insulin Analogs (Insulin Lispro Protamine Suspension and Comparator) in Basal Therapy for Patients With Type 2 Diabetes Mellitus
Brief Title: Comparison of Two Basal Insulins for Patients With Type 2 Diabetes (IOOY)
Acronym: IOOY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10935; F3Z-MC-IOOY
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2009-11-04 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — neutral protamine lispro insulin; Insulin Lispro; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro Protamine Suspension (Experimental): Insulin Lispro Protamine Suspension: Patient specific dose administered subcutaneously once daily or twice daily x 24 weeks.
  Interventions: Drug: Insulin Lispro Protamine Suspension
- Detemir (Active Comparator): Detemir: Patient specific dose administered subcutaneously once or twice daily x 24 weeks.
  Interventions: Drug: Detemir

INTERVENTIONS:
Drug: Insulin Lispro Protamine Suspension — Patient specific dose administered subcutaneously once daily or twice daily x 24 weeks.
  Other Names: Neutral Protamine Lispro (NPL); Humalog; ILPS
  Arms: Insulin Lispro Protamine Suspension
Drug: Detemir — Patient specific dose administered subcutaneously once or twice daily x 24 weeks.
  Arms: Detemir

SUMMARY:
The purpose of this study is to examine the effectiveness and safety of insulin lispro protamine suspension (ILPS) as compared to insulin detemir as basal insulin therapy in adults with type 2 diabetes. A gatekeeper strategy will be employed for sequentially testing the secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Have type 2 diabetes mellitus for at least 1 year.
2. Are at least 18 years old.
3. Have been receiving oral antihyperglycemic medications (OAMs), without insulin, for at least 3 months immediately prior to the study and have been on stable doses of at least 2 of the following OAMs for the 6 weeks prior to Visit 1, at or above the doses defined in the following: Metformin--1500 milligrams per day (mg/day); Sulfonylureas--1/2 the maximum daily dose, according to the local package insert; Dipeptidyl peptidase-intravenous (DPP-IV) inhibitors-- 1/2 the maximum daily dose, according to the local package insert; Thiazolidinediones (TZDs)--30 mg/day pioglitazone or 4 mg/day rosiglitazone.
4. Have a hemoglobin A1c (HbA1c) greater than or equal to 7.5% and less than or equal to 10.0%, as measured by a central laboratory before Visit 2.
5. Body mass index (BMI) greater than or equal to 25 and less than or equal to 45 kilograms per square meter (kg/m2).

Exclusion Criteria

1. Have used insulin therapy (outside of pregnancy) any time in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 weeks.
2. Have taken any glucose-lowering medications not included in Inclusion Criterion [3] (for example, acarbose, miglitol, pramlintide, exenatide, repaglinide, or nateglinide) in the past 3 months before Visit 1.
3. Have had more than 1 episode of severe hypoglycemia, within 6 months prior to entry into the study, or is currently diagnosed as having hypoglycemia unawareness.
4. Have a history of renal transplantation or are currently receiving renal dialysis or creatinine greater than or equal to 2.0 milligrams per deciliter (mg/dL) (177 micromoles per liter [micromol/L]).
5. Have obvious clinical signs or symptoms, or laboratory evidence, of liver disease (alanine transaminase [ALT], or aspartate transaminase [AST] greater than 2 times the upper limit of the reference range, as defined by the local laboratory) or have albumin value above or below the normal reference range, as defined by the local laboratory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (27):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hueytown, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Litchfield Park, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buena Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newburgh, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slidell, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prince Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novi, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goldsboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansdale, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taylors, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Prairie, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menomonee Falls, Wisconsin
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramos Mejía
- Hungary (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eger
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Makó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rzeszów
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sungnam-Si
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lugo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yung-Kang, Tainan

REFERENCES:
- [Derived] Qu Y, Jacober SJ, Zhang Q, Wolka LL, DeVries JH. Rate of hypoglycemia in insulin-treated patients with type 2 diabetes can be predicted from glycemic variability data. Diabetes Technol Ther. 2012 Nov;14(11):1008-12. doi: 10.1089/dia.2012.0099. PMID 23101951
- [Derived] Fogelfeld L, Dharmalingam M, Robling K, Jones C, Swanson D, Jacober S. A randomized, treat-to-target trial comparing insulin lispro protamine suspension and insulin detemir in insulin-naive patients with Type 2 diabetes. Diabet Med. 2010 Feb;27(2):181-8. doi: 10.1111/j.1464-5491.2009.02899.x. PMID 20546262
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 789 patients were screened; 347 patients failed screening or discontinued before randomization. Demographics and outcomes are reported on the "Full Analysis Set": all randomized patients who received at least one dose of study drug and had at least one post-baseline measurement for the dependent variable, according to Intent to Treat principles.
Groups:
- Detemir: Detemir: Patient specific dose administered subcutaneously once daily x 24 weeks.
Period: Overall Study
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Started | 223 | 219
Full Analysis Set (Intent to Treat) | 219 | 210
Completed | 193 | 183
Not Completed | 30 | 36
Not completed — Adverse Event | 0 | 1
Not completed — Entry Criteria Not Met | 1 | 4
Not completed — Lost to Follow-up | 5 | 6
Not completed — Physician Decision | 3 | 5
Not completed — Protocol Violation | 8 | 5
Not completed — Withdrawal by Subject | 13 | 14
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Protamine Suspension | Detemir | Total
Number analyzed (Participants) | 219 | 210 | 429
Age Continuous [Mean (Standard Deviation); unit: years] | 56.32 (9.91) | 55.73 (10.20) | 56.03 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 97 | 205
  Male | 111 | 113 | 224
Region of Enrollment [Number; unit: participants]
  Argentina | 10 | 11 | 21
  Hungary | 36 | 34 | 70
  India | 42 | 39 | 81
  Korea, Republic of | 10 | 11 | 21
  Mexico | 28 | 27 | 55
  Spain | 13 | 13 | 26
  Taiwan | 20 | 19 | 39
  United States | 60 | 56 | 116
Race/Ethnicity [Number; unit: participants]
  African | 8 | 8 | 16
  Caucasian | 88 | 82 | 170
  East Asian | 35 | 33 | 68
  Hispanic | 45 | 47 | 92
  West Asian | 43 | 40 | 83
Sulfonylurea Group [Number; unit: participants] — Patients with previous sulfonylurea use.
  participants
    Yes | 170 | 158 | 328
    No | 49 | 51 | 100
    Unavailable | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilogram per square meter (kg/m^2) | 30.03 (5.01) | 30.10 (5.12) | 30.06 (5.06)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 81.10 (17.46) | 82.72 (19.32) | 81.89 (18.39)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.48 (6.09) | 8.94 (5.59) | 9.22 (5.85)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.94 (10.19) | 165.14 (10.94) | 164.53 (10.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Week Endpoint in Hemoglobin A1c (HbA1c)
Time Frame: Baseline, 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
percent of HbA1c
  Baseline (n=209, n=202) | 8.79 (0.06) | 8.77 (0.06)
  Change from Baseline (n=209, n=202) | -1.52 (0.08) | -1.31 (0.08)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Hypothesis: Basal analog insulin lispro protamine suspension, injected once or twice daily is noninferior to basal analog insulin determir, injected once or twice daily, with regard to glycemic control as measured by change in HbA1c from baseline to endpoint (last observation carried forward); Test type: Non-Inferiority or Equivalence — The noninferiority margin was 0.4%; p = 0.026, ANCOVA; ANCOVA Model: Variable=Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.21, 95% CI [-0.39 to -0.03] — The two-sided 95% confidence interval is for the Least Squares Mean difference between the two treatments (Insulin Lispro Protamine Suspension minus Determir)

2. Secondary Outcome: Actual and Change From Baseline Hemoglobin A1c (HbA1c) Value at 12 Weeks and at 24 Weeks
Time Frame: Baseline, 12 Weeks, 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent hemoglobin
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
percent hemoglobin
  Baseline | 8.79 (0.06) | 8.77 (0.06)
  Week 12 HbA1c | 7.44 (0.08) | 7.55 (0.07)
  Week 12 Change from Baseline | -1.33 (0.08) | -1.22 (0.07)
  Week 24 HbA1c | 7.14 (0.09) | 7.34 (0.08)
  Week 24 Change from Baseline | -1.63 (0.09) | -1.43 (0.08)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.213, ANCOVA — P-value for 12 Week Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.11, 95% CI [-0.28 to 0.06] — The two-sides 95% confidence interval is for the Least Squares Mean difference between the two treatments (Insulin Lispro Protamine Suspension minus Detemir)
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.213, ANCOVA — P-value for 12 Week HbA1c; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.11, 95% CI [-0.28 to 0.06] — The two-sided 95% confidence interval is for the Least Squares Mean difference between the two treatments (Insulin Lispro Protamine Suspension minus Detemir)
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for 24 Week Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.20, 95% CI [-0.38 to -0.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for Week 24 HbA1c; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.20, 95% CI [-0.38 to -0.01] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Percentage of Patients With HbA1c <7.0% and HbA1c < or = 6.5% at Endpoint
Description: Percentage of patients achieving Hemaglobin A1c (HbA1c) targets of less than 7.0% and less than or equal to 6.5% at endpoint.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
percentage of participants
  HbA1c <7.0% | 34.9 | 31.2
  HbA1c ≤6.5% | 22.5 | 16.3
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.463, Fisher Exact — P-value for HbA1c <7.0%
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.135, Fisher Exact — P-value for HbA1c ≤6.5%

4. Secondary Outcome: Glycemic Variability
Description: Glycemic variability was measured by standard deviation (SD) value of fasting blood glucose as measured by intra-patient glycemic variability (determined by the 7-point self-monitoring blood glucose [SMBG] profiles at endpoint) for the actual morning pre-meal blood glucose value.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 218 | 208
millimoles per Liter (mmol/L) | 1.14 (0.64) | 1.04 (0.69)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; The first gatekeeping hypothesis was that Insulin Lispro Protamine Suspension was noninferior to determir; Test type: Non-Inferiority or Equivalence — Noninferiority margin of 0.8 millimoles per Liter (mmol/L); p = 0.107, ANOVA; ANOVA model: Variable=Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group; Mean Difference (Net) = 0.10, 95% CI [-0.02 to 0.23] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: 7-point Self-monitored Blood Glucose (SMBG) Profile at Endpoint
Description: Actual daily mean blood glucose levels at endpoint.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
millimoles per liter (mmol/L)
  Average 7-Point SMBG | 8.25 (1.58) | 8.26 (1.73)
  Average Pre-Meal | 7.48 (1.69) | 7.43 (1.69)
  Average Post-Meal | 9.37 (1.91) | 9.42 (2.21)
  Average Morning+Evening Pre-Meal | 7.49 (1.68) | 7.40 (1.86)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.952, ANOVA — P-value for Average 7-Point SMBG; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.856, ANOVA — P-value for Average Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.790, ANOVA — P-value for Average Post-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.632, ANOVA — P-value for Average Morning+Evening Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group

6. Secondary Outcome: Number of Participants With Self-reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe Hypoglycemia) Overall for All Study Periods
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with: a Roche blood glucose value <2.8 mmol/L or prompt recovery after oral carbohydrate, glucagon, or IV glucose. Results are for the combined titration and maintenance periods.
Time Frame: Baseline to 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
participants
  All Hypoglycemic Episodes | 151 | 137
  Nocturnal Hypoglycemic Episodes | 99 | 68
  Severe Hypoglycemic Episodes (N=214, N=207) | 5 | 2
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.472, Fisher Exact — P-value for All Hypoglycemic Events
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.005, Fisher Exact — P-value for Nocturnal Hypoglycemic Events
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.450, Fisher Exact — P-value for Severe Hypoglycemic Events

7. Secondary Outcome: 1-Year Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe) Overall
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with: a Roche blood glucose value <2.8 mmol/L or prompt recovery after oral carbohydrate, glucagon, or IV glucose. 1-year adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 365.25 days.
Time Frame: Baseline to 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement.
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 1 year
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
hypoglycemic events per 1 year
  Hypoglycemic Rate | 24.23 (32.99) | 16.23 (26.05)
  Nocturnal Hypoglycemic Rate | 6.32 (12.11) | 3.75 (13.18)
  Severe Hypoglycemic Rate | 0.05 (0.45) | 0.01 (0.15)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.001, ANOVA — P-value for Hypoglycemic Rate; Nonparametric ANOVA Model: Rank of Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.001, ANOVA — P-value for Nocturnal Hypoglycemic Rate; Nonparametric ANOVA Model: Rank of Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.226, ANOVA — P-value for Severe Hypoglycemic Rate; Nonparametric ANOVA Model: Rank of Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group

8. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe) Overall
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with: a Roche blood glucose value <2.8 mmol/L or prompt recovery after oral carbohydrate, glucagon, or IV glucose. 30-day adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 30 days.
Time Frame: Baseline to 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement.
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 30 days
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
hypoglycemic events per 30 days
  Hypoglycemic Rate | 1.99 (2.71) | 1.33 (2.14)
  Nocturnal Hypoglycemic Rate | 0.52 (0.99) | 0.31 (1.08)
  Severe Hypoglycemic Rate | 0.00 (0.04) | 0.00 (0.01)

9. Secondary Outcome: Change in Absolute Body Weight (kg) From Baseline to 24 Week Endpoint
Time Frame: Baseline, 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 209
kilograms (kg)
  Baseline | 81.10 (17.46) | 82.56 (19.22)
  Change from Baseline | 1.88 (3.16) | 0.36 (2.85)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; The second gatekeeping hypothesis was that Insulin Lispro Protamine Suspension was noninferior to detemir with regard to change in absolute body weight from baseline to endpoint (last observation carried forward); Test type: Non-Inferiority or Equivalence — Noninferiority margin of 1.5 kilograms (kg); p < 0.001, ANCOVA — P-value for Change from Baseline; ANCOVA Model: Variable=Treatment + Baseline + Country + Baseline HbA1c + Baseline Sulfonylurea Group; Mean Difference (Net) = 1.50, 95% CI [0.93 to 2.06] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Total Daily Insulin Dose (Units) at Endpoint
Description: Insulin dose at endpoint was analyzed by 24-hour total daily insulin (units).
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
Units of insulin | 31.78 (19.14) | 37.30 (29.45)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.074, ANCOVA; ANCOVA Model: Variable=Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group + Change in HbA1c from Baseline

11. Secondary Outcome: Total Daily Insulin Dose Per Body Weight (Units/Kilograms) at Endpoint
Description: Insulin dose at endpoint was analyzed by 24-hour total daily insulin per body weight (Units/kilograms).
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units of Insulin/kilograms (U/kg)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
Units of Insulin/kilograms (U/kg) | 0.39 (0.23) | 0.46 (0.36)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.039, ANCOVA; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Number of Injections of Basal Insulin Analog at Endpoint
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 219 | 210
participants
  Patients with 1 Injection | 89 | 108
  Patients with 2 Injections | 130 | 102
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.026, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Serious Adverse Events (participants affected / at risk) | 7/219 | 1/210
Other Adverse Events (participants affected / at risk) | 78/219 | 70/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Protamine Suspension (N=219) | Detemir (N=210)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro Protamine Suspension (N=219) | Detemir (N=210)
Diabetic retinopathy (Eye disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 7 (7)
Gastritis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (4) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Chest pain (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 3 (3) | 1 (2)
Pain (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3) | 3 (3)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (5)
Nasopharyngitis (Infections and infestations) | 12 (14) | 10 (10)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 7 (8)
Weight increased (Investigations) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 4 (7)
Headache (Nervous system disorders) | 5 (6) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days